CLINICAL TRIAL: NCT01203527
Title: A Study of the Pharmacology of Oseltamivir (Tamiflu-Roche) in Pregnancy
Brief Title: A Study of the Pharmacology of Tamiflu in Pregnancy
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: OPRU Tamiflu
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-08

CONDITIONS: H1N1 Influenza Treatment During Pregnancy
Keywords: H1N1 influenza; Swine flu; Oseltamivir; Tamiflu; Pregnancy
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Tamiflu use during first trimester: This group will consist of twenty-five pregnant women who are being treated with Oseltamivir for clinical indications during the first trimester of their pregnancy.
- Tamiflu use during second trimester: This group will consist of twenty-five pregnant women who are being treated with Oseltamivir for clinical indications during the second trimester of their pregnancy.
- Tamiflu use during third trimester: This group will consist of twenty-five pregnant women who are being treated with Oseltamivir for clinical indications during the first trimester of their pregnancy.
- Tamiflu use in non-pregnant women: This group will consist of twenty-five non-pregnant healthy female volunteers who are being treated with Oseltamivir.

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK) of the anti-flu medication, Tamiflu during pregnancy and to determine to what extent pregnancy may affect the currently recommended dosage of this medication.

DETAILED DESCRIPTION:
The emergence of the novel H1N1 influenza virus has raised concern among public health officials and the public alike. Although initial reports suggested that the risk of serious disease or death was less than initially feared, continued experience suggests that the disease will have a major impact on the public's health. To address this urgent public health challenge, the centers of the Obstetric-Fetal Pharmacology Research Units Network (OPRU) will recruit a total of 75 pregnant women (25 per trimester with singletons pregnancies) who are receiving oseltamivir for supposed influenza infection. When possible, we will recruit women with twin gestation to determine if fetal number affects the drugs pharmacokinetics. We do not anticipated a significant number of multi-fetal gestations (< 10) but even limited data might prove useful in this population given the tremendous change in renal drug clearance that is normally seen in this group of women. An additional 25 healthy non-pregnant women will be studied to define pregnancy- related changes in the PK of oseltamivir and the carboxylate.

We will study each woman once during therapy, performing steady state pharmacokinetic analyses. This study will be performed after 3 days of oral therapy to optimize the possibility that steady state concentrations have been achieved.

We will:

1. collect biological fluids (plasma and urine) to further characterize the pharmacology of the drug;
2. collect a check swab for DNA to allow study of the impact of single nucleotide polymorphisms on drug handing and disease expression;
3. develop an assay or partner with others to develop an assay for oseltamivir and the primary metabolite, oseltamivir carboxylate;
4. compare the pharmacokinetics of oseltamivir and its metabolite in each trimester of pregnancy to evaluate whether gestational age has an impact on the drug's pharmacokinetics;
5. assess the impact of fetal number on the drug's pharmacokinetics;
6. ask all participants about GI tolerance to the drug and any side effects they may be experiencing, especially related to mood and psychiatric well being; and
7. on all pregnant subjects studied, when possible, we will obtain at delivery maternal and umbilical cord blood to evaluate placental transport especially in those who deliver proximate (within 3 days) to drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Taking or about to start oral oseltamivir for presumed influenza viral infection or for prophylaxis
2. Able to give informed consent
3. Pregnant female with singleton or multifetal gestation or healthy non-pregnant female (ancillary study)

Exclusion Criteria:

1. Unable to take medication orally
2. Renal failure - creatinine > 1.5
3. Hct <28

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant and non-pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2007-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Apparent oral clearance of oseltamivir in singletons | At the time of treatment

SECONDARY OUTCOMES:
Apparent oral clearance of oseltamivir in twins | At the time of treatment
Apparent renal clearance of oseltamivir carboxylate in non-pregnant women (ancillary study) | At the time of treatment
Concentration of oseltamivir carboxylate and oseltamivir at times 0 and 12h to ascertain steady state status | At the time of treatment
Plasma esterase activity. (ancillary study) | At the time of treatment
Maternal side effects -GI upset, pregnancy loss, neuropsychiatric disorder | At the time of treatment
Maternal and cord blood oseltamivir and oseltamivir carboxylate concentrations | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beigi, MD, Principal Investigator — University of Pittsburgh; Steve Caritis, MD, Principal Investigator — University of Pittsburgh; Raman Venkataramanan, PhD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington, Seattle, Washington